CLINICAL TRIAL: NCT02335450
Title: Theory Based Intervention Program to Support Physical Activity for Individuals With Multiple Sclerosis: a Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oakland University (Other)
Responsible Party: Principal Investigator, Beth Black, Asst Prof Physical Therapy, Health Sciences, Oakland University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 619511-2
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis
Keywords: exercise; motivational interviewing
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): All five participants in the study will receive this intervention. The participants will be visited in their homes by a physical therapist once a week. The physical therapist will use a coaching technique called motivational interviewing to help the participant develop personal physical activity goals. The participant will discuss their physical activity challenges, and with the help of the physical therapist the participant will set up personal physical activity goals for the following week. The participant will be given a wristband physical activity monitor to wear during the day for four weeks to track their progress in meeting their activity goals.
  Interventions: Behavioral: Motivational Interviewing; Device: Wristband physical activity monitor

INTERVENTIONS:
Behavioral: Motivational Interviewing — The participant will describe their unique physical activity challenges and their physical activity goals with the physical therapist. Using the technique of motivational interviewing, the physical therapist will work with the participant to help identify potential solutions to challenges and set realistic activity goals for the next week. Each week, the participant and the physical therapist will review the previous week's activity data, and the participant's reports of any challenges or problems they encountered in meeting their physical activity goals the previous week. The participant will identify new activity goals for the next week.
  Other Names: Coaching
Device: Wristband physical activity monitor — The participant will wear a Fitbit wristband which will track the participant's daily steps and minutes of physical activity.

SUMMARY:
This study evaluates the effectiveness of personalized physical activity coaching combined with the use of a physical activity monitor to support increased levels of daily physical activity in individuals with multiple sclerosis. All five participants will receive the intervention over the four week intervention phase.

DETAILED DESCRIPTION:
Individuals with multiple sclerosis engage in less daily physical activity than the general population for a variety of reasons. This research project is intended to evaluate whether individualized coaching combined with the use of a Fitbit physical activity wristband monitor will improve physical activity levels in individuals with multiple sclerosis.

Following admission into the study, participants will be visited once a week for four weeks at home by a physical therapist. The participants in consultation with the physical therapist will set daily physical activity goals for the following week and the participants will be taught how to monitor their daily activity using a Fitbit physical activity wristband.

The goals of this study are to determine whether this intervention is effective in helping participants increase their levels of daily physical activity and their confidence that they can successfully engage in daily physical activity. In addition, there will be an evaluation of changes from pre-intervention to post-intervention in quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* must have a physician diagnosis of multiple sclerosis and deemed suitable for engaging in a physical activity program by their physician
* must be ambulatory with or without an assistive device
* must be able to speak and read English
* must have a home computer or device capable of tracking and recording the daily Fitbit physical activity reports

Exclusion Criteria:

* participants will be excluded if any contraindications to engaging in independent exercise are identified during the intake examination by the physical therapist: cardiovascular issues or safety issues with walking.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02-12; Primary Completion 2015-11-12 (Actual); Study Completion 2015-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Black, DSc, Principal Investigator — Oakland University
Locations (1):
- Oakland University, Rochester, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Information will be shared 6 months after publication for one year.
Access Criteria: Principal investigator will consider written request for study protocol and results.

REFERENCES:
- [Background] Borkoles E, Nicholls AR, Bell K, Butterly R, Polman RC. The lived experiences of people diagnosed with multiple sclerosis in relation to exercise. Psychol Health. 2008;23(4):427-41. doi: 10.1080/14768320701205309. PMID 25160577
- [Background] Stroud N, Minahan C, Sabapathy S. The perceived benefits and barriers to exercise participation in persons with multiple sclerosis. Disabil Rehabil. 2009;31(26):2216-22. doi: 10.3109/09638280902980928. PMID 19903131
- [Background] Stroud NM, Minahan CL. The impact of regular physical activity on fatigue, depression and quality of life in persons with multiple sclerosis. Health Qual Life Outcomes. 2009 Jul 20;7:68. doi: 10.1186/1477-7525-7-68. PMID 19619337
- [Background] Rimmer JH, Riley B, Wang E, Rauworth A, Jurkowski J. Physical activity participation among persons with disabilities: barriers and facilitators. Am J Prev Med. 2004 Jun;26(5):419-25. doi: 10.1016/j.amepre.2004.02.002. PMID 15165658
- [Background] Brown C, Kitchen K, Nicoll K. Barriers and facilitators related to participation in aquafitness programs for people with multiple sclerosis: a pilot study. Int J MS Care. 2012 Fall;14(3):132-41. doi: 10.7224/1537-2073-14.3.132. PMID 24453744
- [Background] Motl RW, McAuley E, Sandroff BM. Longitudinal change in physical activity and its correlates in relapsing-remitting multiple sclerosis. Phys Ther. 2013 Aug;93(8):1037-48. doi: 10.2522/ptj.20120479. Epub 2013 Apr 18. PMID 23599354
- [Background] Motl RW, McAuley E, Snook EM. Physical activity and multiple sclerosis: a meta-analysis. Mult Scler. 2005 Aug;11(4):459-63. doi: 10.1191/1352458505ms1188oa. PMID 16042230
- [Background] McGuigan C, Hutchinson M. The multiple sclerosis impact scale (MSIS-29) is a reliable and sensitive measure. J Neurol Neurosurg Psychiatry. 2004 Feb;75(2):266-9. PMID 14742602
- [Background] Rigby SA, Domenech C, Thornton EW, Tedman S, Young CA. Development and validation of a self-efficacy measure for people with multiple sclerosis: the Multiple Sclerosis Self-efficacy Scale. Mult Scler. 2003 Feb;9(1):73-81. doi: 10.1191/1352458503ms870oa. PMID 12617272
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Marcus BH, Selby VC, Niaura RS, Rossi JS. Self-efficacy and the stages of exercise behavior change. Res Q Exerc Sport. 1992 Mar;63(1):60-6. doi: 10.1080/02701367.1992.10607557. PMID 1574662
- [Background] O'Halloran PD, Blackstock F, Shields N, Holland A, Iles R, Kingsley M, Bernhardt J, Lannin N, Morris ME, Taylor NF. Motivational interviewing to increase physical activity in people with chronic health conditions: a systematic review and meta-analysis. Clin Rehabil. 2014 Dec;28(12):1159-71. doi: 10.1177/0269215514536210. Epub 2014 Jun 18. PMID 24942478

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: The participants will be visited in their homes by a physical therapist once a week. The physical therapist will use motivational interviewing to help the participant develop personal physical activity goals. The participant will discuss their physical activity challenges, and with the help of the physical therapist the participant will set up personal physical activity goals for the following week. The participant will be given a wristband physical activity monitor to wear during the day for four weeks to track their progress in meeting their activity goals and keep a daily physical activity log.
Period: Overall Study
Arm/Group | Single Arm
Started | 5
Completed | 4
Not Completed | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: All 5 participants completed baseline questionnaires.
Groups:
- Single Arm: All five participants had multiple sclerosis (MS). Four participants had relapsing-remitting MS and one participant had progressive-relating MS. Years since diagnosis of MS ranged from 9 years to 29 years.
Arm/Group | Single Arm
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 53 [36 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All 5 participants completed baseline questionnaires.
  Participants
    Female | 5
    Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: All 5 participants completed baseline questionnaires.
  participants
    United States | 5
Exercise Self-Efficacy [Mean (Full Range); unit: units on a scale] — The Exercise Self-Efficacy Scale contains 6 statements asking respondents to indicate their level of confidence that they can exercise three times per week for a period of one month, two months, three months, four months, five months and six months. For each of these 6 statements, the respondent selects one answer from 10% increments from 0% to 100%. The responses for all statements are summed and the number is divided by 6.
  The minimum score is 0, the maximum score is 100. Higher values represent a better outcome.
  units on a scale | 72.58 [58.3 to 100.00]
Multiple Sclerosis Impact Scale [Mean (Full Range); unit: units on a scale] — The Multiple Sclerosis Impact Scale (MSIS-29) consists of 29 questions about the impact of multiple sclerosis on the respondent's life during the past two weeks. For each question, the respondent circles the one best number that best describes their situation. The number 1 = Not at all, 2= A little, 3= Moderately, 4= Quite a bit, 5= Extremely. The scores are summed.
  Scores range from 29 to 145. Higher numbers represent a worse outcome.
  units on a scale | 73.8 [37.0 to 109.0]
Multiple Sclerosis Self-Efficacy Scale [Mean (Full Range); unit: units on a scale] — The Multiple Sclerosis Self-Efficacy Scale is a self-report of psychological adjustment and quality of life of individuals with MS. The 14 statements are answered by selecting one of 6 options ranging from strongly disagree to strongly agree. The range of scores is 14 to 84. Higher scores mean better outcomes.
  units on a scale | 51.4 [40.0 to 69.0]

OUTCOME MEASURES:

1. Primary Outcome: Total Steps Taken Over Course of the Study
Description: Wristband physical activity monitor recorded steps taken by participant over the 4 weeks of the study. No minimum or maximum. No baseline taken so cannot compare pre-intervention to post intervention.
Time Frame: 4 weeks
Population: Only 3 of the 4 participants who completed the study were included in the step total. One participant walked too slowly due to her disease to trigger the wristband step monitor.
Measure: Number; unit: steps over 4 weeks
Groups:
- Single Arm: The participants will be visited in their homes by a physical therapist once a week. The physical therapist will use motivational interviewing to help the participant develop personal physical activity goals. The participant will discuss their physical activity challenges, and with the help of the physical therapist the participant will set up personal physical activity goals for the following week. The participant will be given a wristband physical activity monitor and fill out a daily physical activity log to track their progress in meeting their activity goals. Each week, the participant and the physical therapist will review the previous week's activity data, and the participant's reports of any challenges or problems they encountered in meeting their physical activity goals the previous week. The participant will identify new activity goals for the next week.
Arm/Group | Single Arm
Number analyzed (Participants) | 3
steps over 4 weeks | 296,147

2. Secondary Outcome: Exercise Self-Efficacy Questionnaire
Description: The "Exercise Self-Efficacy Scale" is the participant's self-reported confidence in their ability to engage in exercise throughout the day. Each of the 6 items is scored from 0% confidence to 100% confidence. All items are summed and the score is divided by 6 Minimum score: 0 Maximum score:100 Higher scores mean a better outcome.
Time Frame: baseline and at end of 4-week intervention
Population: The 4 participants who completed the study had baseline and end of study exercise self-efficacy measured.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Single Arm Mean Baseline Score; Single Arm Mean Post-study Score: The participants will be visited in their homes by a physical therapist once a week. The physical therapist will use motivational interviewing to help the participant develop personal physical activity goals. The participant will discuss their physical activity challenges, and with the help of the physical therapist the participant will set up personal physical activity goals for the following week. The participant will be given a wristband physical activity monitor to wear during the day for four weeks to track their progress in meeting their activity goals and keep a daily physical activity log.
Arm/Group | Single Arm Mean Baseline Score | Single Arm Mean Post-study Score
Number analyzed (Participants) | 4 | 4
score on a scale | 73.65 [58.30 to 100] | 91.75 [77.00 to 100]

3. Secondary Outcome: Multiple Sclerosis Self-Efficacy Scale
Description: The "Multiple Sclerosis Self-Efficacy Scale" is a self-report of impact of multiple sclerosis on quality of life. The 14 statements are answered by selecting one of six options from strongly disagree to strongly agree.
  Minimum value: 14 Maximum value: 84 Higher scores reflect mean a better outcome.
Time Frame: baseline compared to end of 4-week study
Population: The 4 participants who competed the study had post-study scores compared to baseline scores.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Single Arm Mean Baseline Score; Single Arm Mean Post-study Score: The participants will be visited in their homes by a physical therapist once a week. The physical therapist will use motivational interviewing to help the participant develop personal physical activity goals. The participant will discuss their physical activity challenges, and with the help of the physical therapist the participant will set up personal physical activity goals for the following week. The participant will be given a wristband physical activity monitor and fill out a daily physical activity log to track their progress in meeting their activity goals. Each week, the participant and the physical therapist will review the previous week's activity data, and the participant's reports of any challenges or problems they encountered in meeting their physical activity goals the previous week. The participant will identify new activity goals for the next week.
Arm/Group | Single Arm Mean Baseline Score | Single Arm Mean Post-study Score
Number analyzed (Participants) | 4 | 4
score on a scale | 48.25 [40 to 69] | 47.25 [28 to 66]

4. Secondary Outcome: Multiple Sclerosis Impact Scale
Description: The "Multiple Sclerosis Impact Scale" is a self-report on how multiple sclerosis has impacted day-to-day life during the past 2 weeks. The 29 items are graded by the participants on a 5 point scale rating from "not at all" to "extremely".
  Minimum score: 29 Maximum Score:145 Higher scores mean worse outcome.
Time Frame: baseline compared to end of 4-week study
Population: The 4 participants who completed the study had their end of study score compared to their baseline score.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Single Arm Baseline Mean Score; Single Arm Post-study Mean Score: The participants will be visited in their homes by a physical therapist once a week. The physical therapist will use motivational interviewing to help the participant develop personal physical activity goals. The participant will discuss their physical activity challenges, and with the help of the physical therapist the participant will set up personal physical activity goals for the following week. The participant will be given a wristband physical activity monitor and fill out a daily physical activity log to track their progress in meeting their activity goals. Each week, the participant and the physical therapist will review the previous week's activity data, and the participant's reports of any challenges or problems they encountered in meeting their physical activity goals the previous week. The participant will identify new activity goals for the next week.
Arm/Group | Single Arm Baseline Mean Score | Single Arm Post-study Mean Score
Number analyzed (Participants) | 4 | 4
score on a scale | 78.25 [37 to 109] | 65 [34 to 77]

ADVERSE EVENTS:
Time Frame: 5 weeks
Groups:
- Single Arm: The participants will be visited in their homes by a physical therapist once a week. The physical therapist will use motivational interviewing to help the participant develop personal physical activity goals. The participant will discuss their physical activity challenges, and with the help of the physical therapist the participant will set up personal physical activity goals for the following week. The participant will be given a wristband physical activity monitor to wear during the day for four weeks and maintain a daily physical activity log to track their progress in meeting their activity goals.
  Each week, the participant and the physical therapist will review the previous week's activity data, and the participant's reports of any challenges or problems they encountered in meeting their physical activity goals the previous week. The participant will identify new activity goals for the next week.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
This was a small case series qualitative design study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No